CLINICAL TRIAL: NCT07360223
Title: Internalized Symptoms in Adolescents With Autism Spectrum Disorder (ASD) and Typically Developing Adolescents : Gaining Insight Into Coping Strategies and the Psychological Processes Involved
Status: Not yet recruiting | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: TSA coping
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: ASD coping
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adolescents: Typically developing adolescents (without ASD)
  Interventions: Behavioral: Questionnaire and interview
- Adolescents with autistic traits without a clinical diagnosis of ASD: Adolescents with autistic traits without a clinical diagnosis of ASD: T score between 66-75 on the SRS-2
  Interventions: Behavioral: Questionnaire and interview
- Adolescents diagnosed with ASD: ASD diagnosis made by a specialist physician
  Interventions: Behavioral: Questionnaire and interview

INTERVENTIONS:
Behavioral: Questionnaire and interview — Participants will complete questionnaires and take part in a semi-structured interview

SUMMARY:
Introduction: Adolescents with autism spectrum disorder (ASD) have more mental health problems than typically developping adolescents (without ASD). Coping strategies are a key concern for adolescents with ASD in managing depressive and anxiety symptoms. Currently, few studies have examined the coping strategies used by adolescents with ASD. The methodological considerations underscore the need for an assessment method tailored to adolescents with ASD. Finally, although current data are still limited, the results suggest that there may be differences between the coping strategies used by adolescents with ASD and typically developing adolescents, thus calling for more in-depth comparative research.

Objectives: This study aims to validate a coping strategies assessment method adapted for adolescents with ASD (1) and to examine coping strategies associated with internalizing symptoms (2)

Population: 252 participants: 84 adolescents with ASD (1), 84 adolescents with autistic traits but no clinical diagnosis of ASD (2), and 84 typically developing adolescents (3). The age range is 12-17 years.

Study design: The study is divided into two parts: a cross-sectional part (T) and a longitudinal part (L).

* The cross-sectional part will include three meetings spread over a period of approximately three months (approximately one meeting per month).
* The longitudinal part will consist of a meeting scheduled one year after the last meeting of the cross-sectional part.

ELIGIBILITY:
Inclusion Criteria:

* 12-17 years
* speak french fluently

Exclusion Criteria:

* Intellectual disability

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolescents aged between 12 and 17 with or without ASD
Sampling Method: Non-Probability Sample
Enrollment: 252 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Coping strategies | Throughout the entire study, approximately during 5 years
  Measure by questionnaire and semi-structured interviews. Questionnaire : Coping Strategies Inventory (CSI) The questionnaire is designed to identify coping strategy profiles. It includes 8 sub-strategies (Problem solving, Cognitive restructuring, Express Emotions, Social Support, Problem avoidance, Wishful thinking, Self-Criticism, Social Withdrawal) and does not have strict minimum or maximum scores. Instead, it provides an overview of the relative use of each coping strategy

SECONDARY OUTCOMES:
Anxious, depressive and somatic symptoms | Throughout the entire study, approximately during 5 years
  Measure by questionnaire Questionnaire : Revised Children's Anxiety and Depression Scale (RCADS) T-score < 65 → Non-clinical range. Symptoms are minimal or within the typical range compared to the normative population. No clinical concern is indicated T-score ≥ 65 → Borderline/clinically elevated Symptoms are higher than average and may indicate potential anxiety or depression issues.
  T-score ≥ 70 → Clinically significant range Symptoms are substantially elevated compared to peers. There is a high likelihood of clinically meaningful anxiety or depression

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie NNG Nader-Grosbois, Professor, Principal Investigator — Université Catholique de Louvain (UCLouvain)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rieffe C, Oosterveld P, Terwogt MM, Mootz S, van Leeuwen E, Stockmann L. Emotion regulation and internalizing symptoms in children with autism spectrum disorders. Autism. 2011 Nov;15(6):655-70. doi: 10.1177/1362361310366571. Epub 2011 Jul 6. PMID 21733959
- [Result] Rieffe C, De Bruine M, De Rooij M, Stockmann L. Approach and avoidant emotion regulation prevent depressive symptoms in children with an Autism Spectrum Disorder. Int J Dev Neurosci. 2014 Dec;39:37-43. doi: 10.1016/j.ijdevneu.2014.06.003. Epub 2014 Jun 19. PMID 24951836